CLINICAL TRIAL: NCT02090218
Title: I-Gel Versus Current Practice in Out-of-hospital Cardiac Arrest by Paramedics in Norway - a Prospective Stepped Wedge Crossover Trial
Brief Title: I-Gel in Out-of-hospital Cardiac Arrest in Norway
Acronym: I-CAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients/centres included.
Sponsor: Haukeland University Hospital (Other)
Collaborators: Sykehuset Innlandet HF (Other); Helse Midt-Norge (Other); Helse Fonna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/984/REK-Vest.
Record Dates: First submitted 2014-01-29; First posted 2014-03-18 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2016-06

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-Gel (Active Comparator): I-Gel supraglottic airway device
  Interventions: Device: I-Gel
- LTS, ETI or other airway practice (Active Comparator): Laryngeal tube, endotracheal tube or other current airway management practice
  Interventions: Device: LTS, ETI or current airway management practice

INTERVENTIONS:
Device: I-Gel — I-Gel supraglottic airway device
  Arms: I-Gel
Device: LTS, ETI or current airway management practice — Laryngeal tube, endotracheal tube, bag-mask-ventilation
  Arms: LTS, ETI or other airway practice

SUMMARY:
The main objective of this trial is to compare the effectiveness of a newer supraglottic airway method (the i-Gel), compared to current airway management practice in out-of-hospital cardiac arrests treated by Norwegian ambulance services.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest patients requiring and receiving advanced airway management on ambulance missions. Advanced airway management is defined as the attempted insertion of an airway adjunct (I-Gel, laryngeal tube or ETI) or the administration of ventilatory assistance/support (including bag-mask ventilation (BMV) or other ventilatory support.
* Adult patients (> 18 years).

Exclusion Criteria:

* Non-adult patients / minors (< 18 years).
* Traumatic cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
ventilation success | up to 24 hours
  ventilation success defined as successful insertion of device with visible chest movement with each ventilation, audible air passage on auscultation, and ETCO2 confirmation (if available) of tube placement

SECONDARY OUTCOMES:
survival to hospital discharge / 30-day survival | up to 30 days
levels of ETCO2 related to the presence and quality of bystander CPR | up to 24 hours
cerebral function assessed by Glascow Outcome Score at discharge from hospital | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
insertion related complications | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Geir A Sunde, MD, Principal Investigator — Haukeland University Hospital; Jon-Kenneth Heltne, MD, PhD, Study Chair — Haukeland University Hospital; Guttorm Brattebø, MD, Study Chair — Haukeland University Hospital; Hanne Klausen, MD, Study Director — Haukeland University Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Innlandet Sykehus HF, Brumunddal
  - Helse Fonna HF, Haugesund
  - Ambulanse Midt-Norge HF, Trondheim